CLINICAL TRIAL: NCT06665009
Title: Utilization and Evaluation of Ampoule Peel Device
Brief Title: How Nurses Use and Evaluate the Ampoule Peel Device: Comparing Manually Opened Vs. Device-Opened Ampoules
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chih-Cheng Wu (Other)
Collaborators: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor-Investigator, Chih-Cheng Wu, head, Department of Pain Management, Taichung Veterans General hospital, Taichung Veterans General Hospital
Organization: Taichung Veterans General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CG24481A
Record Dates: First submitted 2024-10-16; First posted 2024-10-30 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Nurse Based Care Management
Keywords: ampoule; ampoule peeling device; Device-Opened Ampoules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Manually Opened and Device-Opened (Experimental)
  Interventions: Device: Manually Opened and Device-Opened Ampoules

INTERVENTIONS:
Device: Manually Opened and Device-Opened Ampoules — this study is to evaluate the ampoule peeling device in terms of safety, ease of use, time efficiency, difficulty of operation, and user satisfaction among nurses when opening ampoule bottles of different capacities

SUMMARY:
Nurses frequently handle ampoule bottles in their daily work, and due to the fragile nature of these glass bottles, manual opening often leads to hand injuries. According to studies, a high proportion of occupational injuries among nurses are caused by handling ampoule bottles, especially hand lacerations. These injuries not only affect work efficiency but also increase medical risks. Therefore, to improve safety and reduce occupational injuries, this study aims to evaluate a patented ampoule peeling device, which has also won the National Innovation Award, to assess whether it can enhance the safety and satisfaction of nurses during their work.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the ampoule peeling device in terms of safety, ease of use, time efficiency, difficulty of operation, and user satisfaction among nurses when opening ampoule bottles of different capacities. A key focus is to determine whether the device can reduce the risk of hand injuries and improve work efficiency.

Study Design and Procedures:

The study will be conducted in three phases:

1. Phase 1 (Experimental Study):

   In a quiet and controlled environment, nurses will manually and using the ampoule peeling device, open different sizes of ampoule bottles (1ml, 2ml, 5ml, 10ml). Each participant will record the time required, safety, difficulty, success rate, and any incidents of hand injuries during the process. After completing both methods, participants will fill out subjective evaluation forms to assess their satisfaction with each method.
2. Phase 2 (Observational Study):

   Nurses participating in Phase 1 will record the number of ampoule bottles they manually open over five consecutive days, noting the success rate and any hand injuries. Then, they will use the ampoule peeling device for the next five days and record similar data for comparison.
3. Phase 3 (Observational Study):

After Phase 2, participants will have the freedom to choose between manual or device-assisted methods for a six-month period. At the end of this period, they will complete a survey summarizing their reasons for choosing a method, usage frequency, and overall safety and satisfaction levels.

Expected Outcomes:

It is anticipated that the ampoule peeling device will significantly improve safety, ease of use, and user satisfaction compared to manual methods. While there may not be a statistically significant difference in time efficiency, the overall success rate and safety should be enhanced.

ELIGIBILITY:
Inclusion Criteria:

* 16 nursing staff members from W72, W75, and the Department of Anesthesiology, who passed the preliminary tests and are willing to continue to the subsequent phases

Exclusion Criteria:

* Nursing staff unwilling to participate, unable to manually break ampoules, experiencing difficulty during the preparatory phase, or deciding to discontinue or withdraw during the process.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-11-29 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
events of injury | through study completion, an average of 1 year
  events times and sites of injury from different volumes of ampoules
time efficiency | through study completion, an average of 1 year
  time spent needed to open ampules manually or by ampoule openers by seconds
subjective estimation of safety | through study completion, an average of 1 year
  subjective estimation of safety by a scale out of a maximum score of 5, with 1 stands for "strongly disagree" and 5 stands for "strongly agree".

SECONDARY OUTCOMES:
ease of use | through study completion, an average of 1 year
  subjective estimation of time-saving and difficulty by a scale out of a maximum score of 5, with 1 stands for "strongly disagree" and 5 stands for "strongly agree"
difficulty of operation | through study completion, an average of 1 year
  subjective estimation of time-saving and difficulty by a scale out of a maximum score of 5, with 1 stands for "strongly disagree" and 5 stands for "strongly agree"
user satisfaction | through study completion, an average of 1 year
  estimation of overall satisfaction rating (Out of a maximum score of 10, with 0 being very dissatisfied and 10 being very satisfied) for either open ampoules manually or by ampoule openers

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan